CLINICAL TRIAL: NCT05791227
Title: EchoNet-LVH-RCT: Blinded, Randomized Controlled Trial of Artificial Intelligence Guided Precision Assessment of Wall Thickness
Brief Title: Safety and Efficacy Study of AI Wall Thickness Measurement (EchoNet-LVH-RCT)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, David Ouyang, Staff Physician, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: STUDY00002521
Record Dates: First submitted 2023-03-03; First posted 2023-03-30 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Studies will be randomized 1:1 to either sonographer preliminary report finding or AI preliminary report finding with final adjudication by the cardiologist. With AI preliminary report, the preliminary interpretations will be generated by AI (artificial intelligence) technology [a semantic segmentation model] and the PACS system's native reporting workflow will be used visualize measurements of left ventricular diameter during diastole (LVIDd), intraventricular septum thickness during diastole (IVSd) and left ventricular posterior wall thickness during diastole (LVPWd). The study team will assess how much cardiologists edit and change this preliminary interpretation is from the final interpretation.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Measurements shown in Picture Archiving and Communication System (PACS) without direct communication between sonographer and cardiologist. Annotations are shown without identifiers on how the annotations were done. Cardiologists are blinded to source of preliminary interpretation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sonographer Annotation (Active Comparator): Currently, sonographer technicians provide preliminary interpretations prior to validation and overreading by cardiologists. This staggered, stepwise evaluation allows for the introduction of AI decision support with minimal impact on patient care. Physicians are already used to adjusting the preliminary report given the variable training of sonographers and on the lookout for changes, variation, or adjustments that need to be made.
  Interventions: Diagnostic Test: Sonographer Evaluation
- Artificial Intelligence Annotation (Experimental): A novel AI algorithm developed to assess measurements of left ventricular diameter during diastole (LVIDd), intraventricular septum thickness during diastole (IVSd) and left ventricular posterior wall thickness during diastole (LVPWd). The AI will provide preliminary assessments for cardiologist evaluation.
  Interventions: Diagnostic Test: AI Evaluation

INTERVENTIONS:
Diagnostic Test: Sonographer Evaluation — A sonographer will assess measurements of left ventricular diameter during diastole (LVIDd), intraventricular septum thickness during diastole (IVSd) and left ventricular posterior wall thickness during diastole (LVPWd).
  Arms: Sonographer Annotation
Diagnostic Test: AI Evaluation — An AI model will assess measurements of left ventricular diameter during diastole (LVIDd), intraventricular septum thickness during diastole (IVSd) and left ventricular posterior wall thickness during diastole (LVPWd).
  Arms: Artificial Intelligence Annotation

SUMMARY:
To determine whether an integrated AI decision support can save time and improve accuracy of assessment of echocardiograms, the investigators are conducting a blinded, randomized controlled study of AI guided measurements of wall thickness in parasternal long axis view compared to sonographer measurements in preliminary readings of echocardiograms.

ELIGIBILITY:
Inclusion Criteria:

* Sonographers and cardiologists at CSMC Echocardiography Lab
* All transthoracic echocardiogram studies performed in the CSMC echocardiogram lab

Exclusion Criteria:

* transthoracic echocardiogram studies not able to be measured by sonographers in run in period

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4000 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of studies for which the difference in wall thickness between preliminary to overread is greater than 0.3cm for LVIDd | 10 Minutes
  Proportion of significant difference in LVIDd between preliminary to final assessment
Proportion of studies for which the difference in wall thickness between preliminary to overread is greater than 0.2cm for IVSd | 10 Minutes
  Proportion of significant difference in IVSd between preliminary to final assessment
Proportion of studies for which the difference in wall thickness between preliminary to overread is greater than 0.2cm for LVPWd | 10 Minutes
  Proportion of significant difference in LVPWd between preliminary to final assessment
mean absolute error (MAE) of LVIDd between preliminary to overread between the two arms | 10 Minutes
  Measurement difference of LVIDd between preliminary to final assessment
mean absolute error (MAE) of IVSd between preliminary to overread between the two arms | 10 Minutes
  Measurement difference of IVSd between preliminary to final assessment
mean absolute error (MAE) of LVPWd between preliminary to overread between the two arms | 10 Minutes
  Measurement difference of LVPWd between preliminary to final assessment

SECONDARY OUTCOMES:
mean absolute error (MAE) of wall thickness between cardiologist overread vs. historical clinical report wall thickness | 10 Minutes
  Mean absolute error (MAE) of wall thickness between cardiologist overread with initial interpretation vs. prior clinical report wall thickness
Time to complete each imaging study | 10 Minutes
  Time for sonographers and cardiologists to complete a study (in seconds)
Effects of the AI systems integration with computer-human interaction (Blinding) | 10 Minutes
  Whether cardiologists can tell the difference between human vs. AI initial interpretation (Bang's blinding index, or the proportion of studies guessed correctly to be AI or sonographer compared to ground truth of whether it was AI or sonographer).

IPD SHARING:
Plan to Share IPD: Undecided